CLINICAL TRIAL: NCT06880926
Title: A Randomized, Double-Blind, Parallel-Controlled, Multicenter Clinical Trial of Antarctic Krill Oil in the Management of Knee Osteoarthritis Pain
Brief Title: Antarctic Krill Oil for Knee Osteoarthritis Pain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KYLL-202412-004-1
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis (OA) of the Knee; Osteoarthritis Knee Pain
MeSH Terms: conditions — Osteoarthritis | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olive oil (Placebo Comparator): Oral administration of olive oil : 2 grams per dose, once daily, for a duration of 24 weeks.
  Interventions: Dietary Supplement: Olive Oil
- Antarctic krill oil (Experimental): Oral administration of antarctic krill oil : 2 grams per dose, once daily, for a duration of 24 weeks.
  Interventions: Drug: Krill oil

INTERVENTIONS:
Drug: Krill oil — Antarctic krill oil was used for intervention in the experimental group.
  Arms: Antarctic krill oil
Dietary Supplement: Olive Oil — Olive oil was used for intervention in the placebo group.
  Arms: Olive oil

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of Antarctic Krill Oil (AKO) as a dietary supplement in managing pain associated with knee osteoarthritis (OA). The main questions it aims to answer are:

①Does AKO reduce daily pain intensity in participants with moderate knee OA?

②What adverse effects do participants experience when taking AKO?

Researchers will conduct a randomized, double-blind study comparing AKO to a placebo (identical appearance without active components) to assess:

* Changes in joint pain severity; ②Functional improvement in daily activities; ③Biochemical safety parameters,etc.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic degenerative disease affecting the entire joint apparatus, characterized by pathological alterations in articular cartilage, subchondral bone, synovium, and joint capsule, clinically manifested by high rates of disability and deformity. With the accelerating aging population in China, the prevalence of OA has risen significantly, garnering substantial academic attention. Current management for early-to-moderate OA predominantly relies on oral non-steroidal anti-inflammatory drugs (NSAIDs), intra-articular hyaluronic acid injections, and glucocorticoids. For advanced cases, total joint arthroplasty remains the definitive intervention, while no disease-modifying therapies have been established to date.

Antarctic krill oil, a nutrient-dense marine extract, contains clinically relevant bioactive components including phospholipids, eicosapentaenoic acid (EPA), and docosahexaenoic acid (DHA), which are critical mediators of its therapeutic potential. Despite emerging interest, clinical evidence regarding krill oil's efficacy in alleviating OA-related pain and improving joint function remains limited, underscoring the need for further exploration of its role in OA management.

This clinical trial aims to evaluate the efficacy and safety of Antarctic krill oil supplementation in reducing pain severity among patients with knee osteoarthritis (KOA), with the ultimate goal of expanding evidence-based therapeutic options for KOA pain management.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-75 years；
* Clinically diagnosed with knee osteoarthritis per the Chinese Guidelines for the Diagnosis and Treatment of Osteoarthritis (2018 edition) issued by the Chinese Medical Association, with Kellgren-Lawrence grade 1-3；
* Knee pain Visual Analog Scale (VAS) score between 4.0 and 8.0；
* Ability to comprehend and complete VAS and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) assessments；
* Willingness and ability to undergo knee MRI examinations.

Exclusion Criteria:

* Ipsilateral hip osteoarthritis;
* Diagnosis of rheumatoid arthritis (RA), ankylosing spondylitis, sarcoidosis, amyloidosis, or any other inflammatory arthritis (e.g., gout, pseudogout);
* Chronic pain syndromes, fibromyalgia, or comorbidities that may confound knee pain assessment;
* Pain intensity in the lower extremities or back equal to or greater than knee pain;
* Arthroscopic or open knee surgery within the preceding 12 months or planned during the study period;
* Oral, intra-articular, or intramuscular corticosteroid use within 6 months prior to screening or during the study;
* Intra-articular hyaluronic acid injection within 6 months prior to screening or during the study;
* High-dose NSAID use (≥ maximum recommended daily dose for osteoarthritis pain relief) within 1 month prior to screening, including but not limited to: Diclofenac ≥150 mg/day; Aceclofenac ≥100 mg/day; Meloxicam ≥15 mg/day; Naproxen ≥1,000 mg/day; Piroxicam ≥20 mg/day; Ibuprofen >2,400 mg/day (Exempt if a ≥4-week washout period is completed prior to Day 1);
* Bleeding disorders or anticoagulant use within 1 month (except low-dose aspirin ≤150 mg/day);
* Regular use of glucosamine, fish oil, or other supplements unless a ≥4-week washout period (≥3 months for fish oil) is completed prior to Day 1;
* Hypersensitivity to trial medications or seafood;
* Administration of any medication within 6 months prior to Day 1 that may interfere with study outcomes, as judged by investigators;
* Pregnancy (positive urine test at screening or Day 1), lactation, or inadequate contraception;
* History of alcoholism, substance abuse, major systemic diseases (e.g., renal, cardiac, hepatic, or gastrointestinal disorders), or conditions deemed by investigators to compromise study participation or data integrity;
* Uncontrolled hypertension (screening blood pressure ≥140/90 mmHg) unless confirmed as non-hypertensive or well-controlled by a specialist;
* Inability to provide informed consent.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale | Baseline and week 24 after treatment initiation
  Joint pain severity was assessed using the Visual Analogue Scale (VAS).
Adverse Reactions | Baseline, weeks 4, 8, 12, 16, 20, and 24 after treatment initiation
  Safety assessment of the treatment requires written documentation of adverse reactions, including their time of occurrence, frequency, and severity grading.
Serious Adverse Reactions | Baseline, weeks 4, 8, 12, 16, 20, and 24 after treatment initiation
  Safety assessment of the treatment requires written documentation of serious adverse reactions, including their time of occurrence, frequency, and severity grading.

SECONDARY OUTCOMES:
WOMAC Pain Subscale | Baseline, weeks 4, 8, 12, 16, 20, and 24 after treatment initiation
  Joint pain severity was assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale.
WOMAC Stiffness Subscale | Baseline, weeks 4, 8, 12, 16, 20, and 24 after treatment initiation
  Degree of joint stiffness was evaluated with the WOMAC Stiffness Subscale.
WOMAC Physical Function Subscale | Baseline, weeks 4, 8, 12, 16, 20, and 24 after treatment initiation
  Joint functional ability was measured by the WOMAC Physical Function Subscale.
Volume of Joint Effusion | Baseline, weeks 12 and 24 after treatment initiation
  To measure the volume of joint effusion, magnetic resonance imaging is used to scan the joint area and calculate the amount of effusion.
VAS Pain Score Change from Baseline | Baseline, weeks 4, 8, 12, 16, 20, and 24 after treatment initiation
  To measure the degree of joint pain, the Pain Visual Analog Scale (VAS) is used for evaluation. The baseline change value of the Pain Visual Analog Scale is obtained by subtracting the initial measurement score at week 0 from the obtained score.

IPD SHARING:
Plan to Share IPD: Undecided